CLINICAL TRIAL: NCT04982770
Title: Medical Triage in a Time of Scarce Resources: a Randomized Controlled Study.
Brief Title: Medical Triage in a Time of Scarce Resources.
Acronym: XPHI-COVID-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: University of Geneva, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1475
Record Dates: First submitted 2021-07-23; First posted 2021-07-29 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2021-10

CONDITIONS: Morals; Covid19; Ethics, Narrative
MeSH Terms: conditions — COVID-19; Narration | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The participants have to read ethical guidelines before they are asked to complete the questionnaire of the Oxford Utilitarianism Scale and exposed to medical triage dilemmas.
  Interventions: Other: Survey
- No intervention (No Intervention): The participants do not have to read ethical guidelines before they are asked to complete the questionnaire of the Oxford Utilitarianism Scale and exposed to medical triage dilemmas.

INTERVENTIONS:
Other: Survey — Reading of ethical guidelines.
  Arms: Intervention

SUMMARY:
The XPHI-COVID-2 randomized study aims to investigate the moral choices in a context of scarce resources.

The participants are asked to complete the questionnaire of the Oxford Utilitarianism Scale and are exposed to medical triage dilemmas.

Participants are randomized between a group with reading of ethical guidelines and a group without reading of ethical guidelines, before they are asked to complete the questionnaire and being exposed to triage dilemmas.

DETAILED DESCRIPTION:
It is hypothesized that recalling ethical values before resolving dilemmas could modify the ability to adopt a utilitarian approach in resolving ethical dilemmas.

To verify this hypothesis, the score on the Impartial Harm subscale of the Oxford Utilitarianism Scale (IH-OUS) will be compared between a group with reading of ethical guidelines and a group without reading of ethical guidelines, before they are asked to complete the questionnaire and being exposed to triage dilemmas.

Number of subjects needed for the phase of study evaluating intensivists, anesthesiologists and emergency physicians : 580 - based on preliminary data, assuming 70% complete response rate of the survey and a standard deviation of 5

Secondary outcomes will be considered :

* Beneficence Harm subscale of the Oxford Utilitarianism Scale (IB-OUS)
* Values prioritized to resolve ethical dilemmas : impartial of benefits, prioritization of the young age, saving life years, saving most lives, equality of treatment, prioritization of the worst off, loyalty duty, principle of non-discrimination, prospective and retrospective instrumental value.

First phase of the study will aim to include first-line caregivers : intensivists, anesthesiologists, emergency physicians.

Other phases of the study will aim to include health care professionals from other categories and non health care professionals.

Subgroup analyses are planned :

* Analysis according to the characteristics of the participant: gender, geographic location, diploma and type of exercise, category of institution to which the participant is attached.
* Analysis according to the degree of knowledge in ethics, the degree of familiarity with ethical recommendations, the degree of familiarity with moral philosophy, the degree of religiosity, whether the participants declare to have taken knowledge or not of recommendations concerning medical triage in a situation of scarce resources.

It is also planned to carry out ancillary studies in parallel with the realization of the study presented here:

* A study including non-physician participants aiming to identify the differences between non-physicians and physicians in terms of ethical values mobilized in medical triage.
* A study including medical students aiming to identify an association between propensity to make utilitarian and choices of the medical specialty.
* A study focused on the Oxford Utilitarianism Scale, integrating the results of the pilot study and the confirmatory study, aiming to identify predictors of responses to the dilemmas proposed within the scale.
* A study evaluating the association between delay in ethical dilemmas resolution and utilitarian choices.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers
* Noncaregivers from general population

Exclusion Criteria:

* Withdrawal of agreement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
IH-OUS score | At the end of the inclusion period
  Score on the Impartial Harm subscale of the Oxford Utilitarianism Scale (IH-OUS) : minimum value is 4 points and maximum value is 28 points.
  The higher the value is, the more the participant's choices endorse the principle of causing harm to bring the greater good.

SECONDARY OUTCOMES:
Utilitarian score | At the end of the inclusion period
  One point is given for each choice consistent with utilitarian principles when solving triage dilemmas, scaling this score from 0 to 14.
IB-OUS score | At the end of the inclusion period
  Score on the Instrumental Beneficence subscale of the Oxford Utilitarianism Scale (IB-OUS) : minimum value is 5 points and maximum value is 35 points.
  The higher the value is, the more the participant's choices endorse the impartial maximization of the greater good, even at the cost of personal self-sacrifice.
Oxford utilitarianism scale | At the end of the inclusion period
  Bi-dimensional scale of utilitarian thinking associating the impartial harm and the beneficence subscale. The minimum value is 9 points and the maximum value is 63 points.
  This scale aims to assess the utilitarian tendencies in people who are not philosophy professionals.
Impartial of benefits | At the end of the inclusion period
  Principle of impartial assignment of resources used in resolving ethical dilemmas.
  The value will be considered as respected by the majority of participants if more than 50% of respondents make a choice of a patient in accordance with this value.
Prioritization of the young age | At the end of the inclusion period
  Propensity to prioritize the youngest person in ethical dilemmas. The value will be considered as respected by the majority of participants if more than 50% of respondents make a choice of a patient in accordance with this value.
Saving life years | At the end of the inclusion period
  Propensity to save the most life years in resolving ethical dilemmas. The value will be considered as respected by the majority of participants if more than 50% of respondents make a choice of a patient in accordance with this value.
Saving most lives | At the end of the inclusion period
  Propensity to save most lives in resolving ethical dilemmas. The value will be considered as respected by the majority of participants if more than 50% of respondents make a choice of a patient in accordance with this value.
Equality of treatment | At the end of the inclusion period
  Propensity to treat people equally in ethical dilemmas. The value will be considered as respected by the majority of participants if more than 50% of respondents make a choice of a patient in accordance with this value.
Prioritization of the worst off | At the end of the inclusion period
  Propensity to prioritize the worst off in ethical dilemmas. The value will be considered as respected by the majority of participants if more than 50% of respondents make a choice of a patient in accordance with this value.
Duty of loyalty | At the end of the inclusion period
  Propensity of the caregiver to feel obliged vis-a-vis the patient The value will be considered as respected by the majority of participants if more than 50% of respondents make a choice of a patient in accordance with this value.
Principle of non-discrimination (based on age, disability, socio-economic characteristics, gender, etc.) | At the end of the inclusion period
  The non-discrimination principle requires the equal treatment of an individual or group irrespective of their particular characteristics.
  The value will be considered as respected by the majority of participants if more than 50% of respondents make a choice of a patient in accordance with this value.
Prospective instrumental value | At the end of the inclusion period
  Propensity to promote and reward prospective instrumental value, based on future facts.
  The value will be considered as respected by the majority of participants if more than 50% of respondents make a choice of a patient in accordance with this value.
Retrospective instrumental value | At the end of the inclusion period
  Propensity to promote and reward retrospective instrumental value, based on past facts.
  The value will be considered as respected by the majority of participants if more than 50% of respondents make a choice of a patient in accordance with this value.

CONTACTS AND LOCATIONS:
Overall Officials: Clément GAKUBA, MD PhD, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, Calvados, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kahane G, Everett JAC, Earp BD, Caviola L, Faber NS, Crockett MJ, Savulescu J. Beyond sacrificial harm: A two-dimensional model of utilitarian psychology. Psychol Rev. 2018 Mar;125(2):131-164. doi: 10.1037/rev0000093. Epub 2017 Dec 21. PMID 29265854
- [Background] Capraro, V., Earp, B.D., & Everett, J.A.C. (2019). Priming intuition disfavors instrumental harm but not impartial beneficence. Journal of Experimental Social Psychology. 83, 142-149. DOI: 10.1016/j.jesp.2019.04.006.
- [Background] Emanuel EJ, Persad G, Upshur R, Thome B, Parker M, Glickman A, Zhang C, Boyle C, Smith M, Phillips JP. Fair Allocation of Scarce Medical Resources in the Time of Covid-19. N Engl J Med. 2020 May 21;382(21):2049-2055. doi: 10.1056/NEJMsb2005114. Epub 2020 Mar 23. No abstract available. PMID 32202722